CLINICAL TRIAL: NCT01300299
Title: STEREOtactic Radiation and Adjuvant Chemotherapy in Lung Cancer (STEREO)
Brief Title: STEREOtactic Radiation and Chemotherapy in Lung Cancer (STEREO)
Acronym: STEREO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-LUN-10-STEREO
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: lung cancer; radiation; stereotactic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): Subjects will receive chemotherapy after stereotactic body radiation therapy.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — 12 Gray (Gy) x 4 fractions (48 Gy) will be delivered to peripherally located tumors (> 2 cm in all directions around the proximal bronchial tree and centrally located tumors (within <2 centimeters (cm) of proximal bronchial tree). Treatment should be given on consecutive days. There will be 4 or 5 treatments.

SUMMARY:
This trial will test the feasibility of adjuvant chemotherapy after stereotactic body radiation therapy for early stage non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study evaluates the effect of adjuvant chemotherapy in patients who received treatment with stereotactic radiation for early stage lung cancer and who are at high risk for microscopic metastatic disease.

Chemotherapy in the form of cisplatin/docetaxel or cisplatin/pemetrexed will be administered approximately six weeks after Stereotactic Body Radiation Therapy (SBRT). Patients will then undergo follow up clinical evaluation and imaging to evaluate treatment response and for surveillance.

A patient population of 65 patients will be required. Enrollment in this protocol is planned by multi center involvement in the state of Kentucky as part of the Kentucky Trial Network (KTN).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Histologically diagnosed non-small cell lung cancer(NSCLC, cT1-T3 (<= 5cm) (AJCC 7ed). The following histologies are eligible: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, large cell neuroendocrine, or non-small cell carcinoma not otherwise specified; bronchioloalveolar cell carcinoma is a subtype of NSCLC but will be excluded from this study because assessment of multifocal disease spread through the airways is difficult.
* Required CT of the chest and abdomen with contrast unless medically contraindicated (evaluating both lungs, mediastinum, liver, and adrenals) and Whole Body Positron Emission Tomography (PET) for staging. An integrated PET/Computed Tomography (CT) will meet the CT and PET requirements for staging. Images must be read by a trained radiologist and performed 8 weeks prior to initiation of treatment. PET imaging must allow adequate visualization of the primary tumor, draining lymphatics in hilar and mediastinum, adrenals, and skeleton.

Note: Per Radiation Therapy Oncology Group (RTOG) 0915 inclusion criteria, patients with hilar or mediastinal lymph nodes ≤ 1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer.

* Deemed medically inoperable by an experienced thoracic cancer clinician for a standard lobectomy and lymph node sampling/dissection. Inoperability may be defined utilizing a number of criteria. These include any of the following:
* Pretreatment Forced Expiratory Volume (FEV1) < 40% predicted
* Postoperative FEV1 < 30% predicted
* Severely reduced diffusion capacity
* Baseline hypoxemia and/or hypercapnia
* Exercise oxygen consumption < 50% predicted
* Severe pulmonary hypertension
* Diabetes mellitus with severe end organ damage
* Severe cerebral, cardiac, or peripheral vascular disease
* Decline surgery after evaluation by a thoracic surgeon

Required laboratory values within 2 weeks of chemotherapy initiation

* Absolute neutrophil count (ANC) ≥ 1500 mm3
* Platelets ≥ 100,000/mm3
* Total Bilirubin ≤ 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT)- aspartate aminotransferase (AST) < 5 x upper limit of normal (ULN}
* Serum glutamic pyruvic transaminase (SGPT)- alanine transaminase(ALT) < 5 x upper limit of normal (ULN)
* Serum Creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
* For patients assigned to pemetrexed/Cisplatin therapy calculated Creatinine Clearance (CrCl) must be obtained within 2 weeks of randomization and calculated CrCl must be > 45mL/min using the standard Cockcroft and Gault formula

Exclusion Criteria:

* Primary lesion size not within the acceptable criteria
* Evidence of regional metastases or distant metastases following appropriate staging
* Previous radiation to the chest
* Chemotherapy within the previous five years
* Previous surgery for this particular lung tumor
* Plans for concomitant chemotherapy with radiation
* Active systemic or pulmonary infection
* Pregnant or lactating females
* Synchronous primary malignancy or prior malignancy in the past 2 years except for invasive malignancy that has been treated definitively and the patient remains disease free for > 3 years with life expectancy > 3 years. Previous skin cancers and carcinoma in situ treated definitively are acceptable.
* Patients assigned to pemetrexed/cisplatin therapy must NOT have squamous cell histology
* Bronchioloalveolar cell carcinoma is excluded because assessment of multifocal disease spread through the airways is difficult
* Receipt of any other investigational agents or participation in any other investigational drug study within 4 weeks preceding initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To measure the feasibility of adjuvant chemotherapy after stereotactic body radiation therapy for early stage non-small cell lung cancer (NSCLC) | 3 years after subject enrollment

SECONDARY OUTCOMES:
Survival rate, specifically disease-free survival (DFS) and overall survival (OS), measured by follow-up visits and tests | 3 years after subject enrollment
safety of adjuvant chemotherapy after stereotactic body radiation therapy for early stage non-small cell lung cancer (NSCLC) measured by adverse events | 3 years after subject enrollment
quality of life (QOL) measured by subject questionnaires | 3 years after subject enrollment
Measurement of biological and clinical markers for toxicity, DFS, and OS | 3 years after subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States